CLINICAL TRIAL: NCT05147480
Title: The Effects of Online Mother-Baby Yoga on Preterm Infants and Their Mothers
Brief Title: Online Mother-Baby Yoga With Preterm Infants and Their Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Online Mother-Baby Yoga
Record Dates: First submitted 2021-11-15; First posted 2021-12-07 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Preterm Birth; Anxiety; Development, Infant
Keywords: premature infants; yoga; motor performance; COVID-19
MeSH Terms: conditions — Premature Birth; Anxiety Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: Intervention group (yoga) and control group (standardized protocol)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga group (Active Comparator): infants whose gestational ages are between 32-37 weeks and completed the corrected age of the 6th week, and their mothers intervention: 6-week, once a week internet-based mother and baby yoga
  Interventions: Other: internet-based mother-baby yoga
- control group (No Intervention): infants whose gestational ages are between 32-37 weeks and completed the corrected age of the 6th week, and their mothers the standardized follow-up without intervention

INTERVENTIONS:
Other: internet-based mother-baby yoga — Mother-baby yoga group classes given by physiotherapists via Zoom Video Communications
  Arms: yoga group

SUMMARY:
The purpose of this study is to examine the effects of internet-based mother-baby yoga on preterm infants and their mothers.

DETAILED DESCRIPTION:
Mother-infant pairs were enrolled in the study. Interventions applied as group sessions (maximum of 5 mother-infant pairs) for 6 weeks, once a week. Yoga sessions Before-after evaluations were done for both mother and infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The infants whose gestational age between 32 0/7-36 6/7 week and corrected age's older than 6 weeks and their mothers
* Caregivers who have at least one smartphone or/and laptop or/and Ipad
* Mothers and their babies who accept to register to the study

Exclusion Criteria:

* The infants who have a severe pathological sign in cranial screening
* The infants who had IVH
* The infants who have congenital abnormalities
* The infants who have a metabolic or genetic diagnosis
* The infants who have hearing or visual impairment
* The mothers who had chronic depression history and/or mental retardation
* The mothers who have a neurological or orthopedic diagnosis to the contraindication of exercise
* The mothers who are pregnant

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Motor performance of infants | 15 minutes
  Alberta Infant Motor Scale (AIMS)

SECONDARY OUTCOMES:
Anxiety levels of mothers | 15 minutes
  State-Trate Anxiety Inventory (STAI)
Postpartum bonding of mothers | 15 minutes
  Postpartum Bonding Questionnaire (PPBQ)
Nordic Musculoskeletal Questionnaire (NMQ) | 10 minutes
  Musculoskeletal problems of mothers
Health-related quality of life of mothers | 15 minutes
  World health organization quality of life questionnaire (WHOQOL-BREF-TR)

CONTACTS AND LOCATIONS:
Overall Officials: dilara bozgan, Study Director — Istanbul University; mine çalışkan, Prof.Dr., Principal Investigator — Istanbul University
Locations (1):
- Dilara Bozgan, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Bozgan-Bas D, Ince EZ, Kavram G, Caliskan MM. Tele-MiYo: A tele-yoga program for mother-preterm infant dyads. J Bodyw Mov Ther. 2025 Jun;42:192-197. doi: 10.1016/j.jbmt.2024.12.018. Epub 2024 Dec 12. PMID 40325668